CLINICAL TRIAL: NCT03586115
Title: Evaluation of Minimal Hepatic Encephalopathy by a Neurophysiological Test in Patients With Hereditary Hemorrhagic Telangiectasia
Brief Title: Minimal Hepatic Encephalopathy in Hereditary Hemorrhagic Telangiectasian
Acronym: mHE-HHT
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Clinical professor, University of Bari
Other Study IDs: Policlinic Hospital 4, Bari
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hepatic Encephalopathy; Minimal Brain Dysfunction
MeSH Terms: conditions — Hepatic Encephalopathy; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hereditary telangectasia: In addition to all laboratory analyses and imaging studies required to evaluate the disease, hepatic elastometry and critical flicker frequency assessment will be performed.
  Interventions: Device: Critical flicker frequency assessment

INTERVENTIONS:
Device: Critical flicker frequency assessment — All patients will undergo critical flicker frequency assessment to evaluate the presence of minimal hepatic encephalopaty. In addition, hepatic elastometry will be assessed to evaluate the presence of advanced liver fibrosis.
  Other Names: Hepatic elastometry

SUMMARY:
HHT or Rendu-Osler-Weber disease is a genetic disease with an autosomal dominant inheritance pattern, characterized by widespread telangiectases that can involve several organs including the intestinal tract and the liver. Liver involvement by HHT is characterized by widespread diffuse liver vascular malformations that give origin to arteriovenous, arterioportal and portovenous shunts. The prevalence of hepatic involvement in HHT can reach 78%. Less commonly, patients may also develop porto-systemic encephalopathy (PSE). However, there are no studies on the possibility that patients with HHT might develop mHE, a highly plausible hypothesis considering the presence of diffuse macroscopic and microscopic porto-systemic shunt in this pathological condition.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a potentially reversible disorder characterized by neuropsychiatric abnormalities and motor disturbances that range from mild alterations of cognitive and motor functions to coma and death (1-2). This condition has been linked to the combination of gut flora alterations, which increase the production of gut-derived toxins such as ammonia and indoles, and porto-systemic shunts, leading to endotoxemia associated to systemic and cerebral inflammation (3-4). The subclinical expression of HE is defined minimal hepatic encephalopathy (mHE) (5-7). The latter condition is characterized by the presence of various quantifiable neurophysiological and neuropsychological deficits that are only recognized by the use of specific diagnostic tools such as the paper-and-pencil tests and its variants as well as critical flicker frequency (CFF) (8-11).

The visual test based on CFF measures the frequency (Hz) when impression of fused light turns to a flickering one (5,11). This neurophysiological test has an elevated specificity and reproducibility, with only little biases due to training effects and daytime variability (7,11-13). CFF has also shown the ability to predict the risk of developing overt HE in cirrhotics undergoing transjugular intrahepatic portosystemic shunt (TIPS) (14,15).

HHT or Rendu-Osler-Weber disease is a genetic disease with an autosomal dominant inheritance pattern, characterized by widespread telangiectases that can involve several organs including the intestinal tract and the liver (16). There are two main types of the disease, HHT1 and HHT2, which are caused respectively by mutations in ENG gene on chromosome 9 coding for endoglin for HHT1and mutations in ACVRL1 gene on chromosome 12 for HHT2 (17,18). These two types of the disease account for most clinical cases but mutations in MADH4 gene on chromosome 5 (encodingSMAD4), have been recently described, and a new type HHT3 has been reported (17). HHT2 is associated with a high rate of liver involvement (18).

Liver involvement by HHT is characterized by widespread diffuse liver vascular malformations that give origin to arteriovenous, arterioportal and portovenous shunts. The prevalence of hepatic involvement in HHT can reach 78% (19). Less commonly, patients may also develop porto-systemic encephalopathy (PSE) (20). However, there are no studies on the possibility that patients with HHT might develop mHE, a highly plausible hypothesis considering the presence of diffuse macroscopic and microscopic porto-systemic shunt in this pathological condition.

ELIGIBILITY:
Inclusion Criteria:

* In this study all patients with hereditary hemorragic telangectasia carrying micro or macro porto-systemic vascular shunts will be enrolled.

Exclusion Criteria:

* Actual or previous presence of overt HE (West-Haven criteria) (1,2), gastrointestinal bleeding in the previous 2 weeks, significant comorbidities such as cardiac, respiratory or renal failure; previous transjugular intrahepatic portosystemic shunt, electrolyte imbalance as hyponatremia (Na<125 mg/dl), neurological diseases, color blindness or severe visual disturbances (cataracts, diabetic retinopathy), hepatocellular carcinoma or other malignancies, use of psychotropic drugs in the week prior to the study. Patients with advanced liver disease will also be excluded. Diagnosis of cirrhosis or advanced liver fibrosis will be based on: a) histological evaluation documented at any time before enrollment, b) liver transient elastography and c) a combination of clinical, laboratory and abdominal ultrasound parameters established a priori (Barone M et al. Digestive and Liver Disease 2018;50:496-500).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis of hereditary hemorragic telangectasia carrying micro or macro porto-systemic vascular shunts
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Minimal hepatic encephalopaty | one day
  This condition is not clinically evident and therefore it requires specific diagnostic tools (hepatonorm device: measures the critical flicker frequency; the measurement is expressed by Hz) to be diagnosed

SECONDARY OUTCOMES:
Liver fibrosis | one day
  The presence of advanced fibrosis can suggest the development of cirrhosis. Fibrosis is measured by hepatic elastometry and is expressed by kPa

CONTACTS AND LOCATIONS:
Overall Officials: michele barone, MD, PhD, Principal Investigator — University of Bari
Locations (1):
- Policlinic Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barone M, Shahini E, Iannone A, Viggiani MT, Corvace V, Principi M, Di Leo A. Critical flicker frequency test predicts overt hepatic encephalopathy and survival in patients with liver cirrhosis. Dig Liver Dis. 2018 May;50(5):496-500. doi: 10.1016/j.dld.2018.01.133. Epub 2018 Jan 31. PMID 29530628